CLINICAL TRIAL: NCT04793555
Title: Validation of an Apartment to Monitor Human Behaviour During Day and Night
Brief Title: Validation of the NeuroTec Loft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: NLoft_H_1
Record Dates: First submitted 2021-03-03; First posted 2021-03-11 (Actual); Last update posted 2022-08-11 (Actual); Status verified 2022-08

CONDITIONS: Neurodegenerative Diseases; Activities of Daily Living; Aging
MeSH Terms: conditions — Neurodegenerative Diseases

STUDY DESIGN:
Intervention Model Description: Single-center prospective non-inferiority study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental_Arm (Experimental): Assessment of behavior during day and night by unobtrusive sensors
  Interventions: Other: Monitoring by unobtrusive sensors

INTERVENTIONS:
Other: Monitoring by unobtrusive sensors — During the study the behavior of daily activities will be monitored by unobstructive sensors. Most of the sensors will be mounted on the wall or on furniture with direct sight to the participant and thus will not have any physical contact, except some wearables during the stay in the apartment and at home (e.g. watch, mobile polysomnography).

SUMMARY:
The progression of neurodegenerative disorders and the increasing number of elderly people intensifies the need of institutional care, which contrasts with the desire of most elderly and patients to live independently at home. The rapid evolution of assistive technology offers new possibilities in providing medical professionals preventive services in real-time. Therefore, the main focus of this study is on the individual sensors and how they can be combined to one unobtrusive system to assess the human behaviour and daily activities during day and night in an instrumented apartment in healthy participants.

DETAILED DESCRIPTION:
The higher prevalence of age-associated neurodegenerative disorders (e.g. Parkinson, Alzheimer), is in line with a steady increase of the average life expectancy in Switzerland. With the progression of neurodegenerative disorders and the increasing number of elderly people, the need for institutional care intensifies, which contrasts with the desire of most elderly and patients to live independently. The rapid evolution of assistive technology offers new possibilities in providing medical professionals preventive services in real-time. An extended stay in the hospital could influence independent ageing negatively and thus, monitoring has great potential to prevent critical events. In this study, the main focus is on the individual sensors and how they can be combined to one unobtrusive system. In addition, to get an understanding which parameters of the sensors are important and how the data can be extracted and processed (algorithms). Therefore, the aim of this study is to validate the accuracy to assess human behaviour and daily activities during day and night by unobtrusive sensors in an instrumented apartment in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Aged ≥18 years
* German speaking

Exclusion Criteria:

* Infected by multidrug-resistant bacteria according to current medical history
* Incontinence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
Heart rate (Vital parameters) | 1 Week / Continuously
  The heart rate will be continuously measured by pressure sensors, radar sensors, infrared camera, galvanic sensor and polysomnography (gold standard).
Respiration rate (Vital parameters) | 1 Week / Continuously
  The respiration rate will be continuously measured by pressure sensors, radar sensors, infrared camera, galvanic sensor and polysomnography (gold standard).
Oxygen saturation (Vital parameters) | 1 Week / Continuously
  The oxygen saturation will be continuously measured by pressure sensors, radar sensors, infrared camera, galvanic sensor and polysomnography (gold standard).
Systolic / Diastolic blood pressure (Vital parameters) | 1 Week / Continuously
  The blood pressure will be continuously measured by pressure sensors, radar sensors, infrared camera, galvanic sensor and polysomnography (gold standard).
Skin conductance (Vital parameters) | 1 Week / Continuously
  The skin conductance will be continuously measured by pressure sensors, radar sensors, infrared camera, galvanic sensor and polysomnography (gold standard).

SECONDARY OUTCOMES:
3D Model (Coordinates of the joints over time) of the participant in the apartment (Movement parameters) | 1 Week / Continuously
  The pose will be assessed continuously by pressure sensors, radar sensors, accelerometer, gyroscope, motion tracking (gold standard), lidar sensors, piir sensors.

OTHER OUTCOMES:
Usability | Each day / 7x
  The usability of the sensor system will be assessed by the System usability scale (SUS). The score range is between 0 and 100, whereas the higher score means higher usability.
Doors open and closed (Activities of daily living) | 1 Week / Continuously
  Unit: 1 open, 0 closed.
Power used - Power Plugs (Activities of daily living) | 1 Week / Continuously
  Unit: Watt.
Temperature (Activities of daily living) | 1 Week / Continuously
  Unit: Degree Celsius.
Relative Humidity (Activities of daily living) | 1 Week / Continuously
  Unit: Percent - Relative to a maximum humidity given the same temperature.
Brightness (Activities of daily living) | 1 Week / Continuously
  Unit: Lux.
Accelerometer - Wearable (Activities of daily living) | 1 Week / Continuously
  Unit: m/s^2.
Electrocardiography (ECG) - Wearable (Activities of daily living) | 1 Week / Continuously
  Unit: Component of the ECG (QRS Complex).
Cognition 1 | Measured on the first day / 1x
  Cognition will be assessed by the Montreal Cognitive Assessment (MoCA). Scores of the MoCA range from 0 to 30, with a score of 26 and higher generally considered normal.
Cognition 2 | Measured on the first day / 1x
  Cognition will be assessed by the Mini-Mental State Examination (MMSE). Scores of the MMSE range from 0 to 30, with a score of 25 and higher generally considered normal.
Health-related quality of life | Measured on the first and last day / 2x
  Health-related quality of life will be assessed by the EuroQol (EQ-5D-5L).The EQ-5D-5L comprises five questions on mobility, self-care, pain, usual activities, and psychological status. The questions have five possible answers for each item (no problems - unable to).
Sleep quality | Each day / 7x
  Sleep quality will be assessed by the SF A/R. The inventory estimates the total sleep duration (calculated from items 'bedtime in the evening' and 'wake-up time in morning'), time awake after sleep onset, and sleep onset latency (5-point Likert scale).
Chronotype | Measured on the first day / 1x
  The Chronotype will be assessed by the D-MEQ. The D-MEQ scores range between 13 and 86. High sum scores (59-86) are associated to morningness, while lower scores point to eveningness (16-41).
Depression 1 | Measured on the first day / 1x
  Depression will be assessed by the Geriatric Depression Scale (GDS). The inventory has 15 questions (yes/no). Scores of 0-4 are considered normal and 12-15 indicate severe depression.
Depression 2 | Measured on the first day / 1x
  Depression will be assessed by the Beck Depression Inventory (BDI). The inventory has 21 questions (yes/no). Scores of 1-10 are considered normal and over 40 indicate severe depression.
Physical activity | Measured on the first day / 1x
  Physical activity will be assessed by the International Physical Activity Questionnaire (IPAQ). The IPAQ assesses the time spent on walking, doing moderate-intensity and vigorous-intensity activity within the domains of work, transportation, domestic and gardening (yard) activities, and leisure-related activities.
Grip strength | Measured on the first day / 1x
  Grip strength will be assessed by a dynamometer.
Fall risk | Measured on the first day / 1x
  Fall risk will be assessed by the Time Up and Go Test (TUG).
Gait and balance | Measured on the first day / 1x
  Gait and balance will be assessed by the Tinetti Balance and Gait Test (POMA).

CONTACTS AND LOCATIONS:
Overall Officials: Stephan M Gerber, PhD, Principal Investigator — Gerontechnology & Rehabilitation Group, University of Bern, Switzerland
Locations (1):
- ARTORG Center for Biomedical Engineering, Gerontechnology and Rehabilitation, Bern, Ber, Switzerland

IPD SHARING:
Plan to Share IPD: No
Data will be available after the publication of the results upon request.

REFERENCES:
- [Background] Andersen CK, Wittrup-Jensen KU, Lolk A, Andersen K, Kragh-Sorensen P. Ability to perform activities of daily living is the main factor affecting quality of life in patients with dementia. Health Qual Life Outcomes. 2004 Sep 21;2:52. doi: 10.1186/1477-7525-2-52. PMID 15383148
- [Background] Saner H, Schutz N, Botros A, Urwyler P, Buluschek P, du Pasquier G, Nef T. Potential of Ambient Sensor Systems for Early Detection of Health Problems in Older Adults. Front Cardiovasc Med. 2020 Jul 15;7:110. doi: 10.3389/fcvm.2020.00110. eCollection 2020. PMID 32760739
- [Background] Schutz N, Saner H, Rudin B, Botros A, Pais B, Santschi V, Buluschek P, Gatica-Perez D, Urwyler P, Marchal-Crespo L, Muri RM, Nef T. Validity of pervasive computing based continuous physical activity assessment in community-dwelling old and oldest-old. Sci Rep. 2019 Jul 4;9(1):9662. doi: 10.1038/s41598-019-45733-8. PMID 31273234
- [Background] Urwyler P, Stucki R, Rampa L, Muri R, Mosimann UP, Nef T. Cognitive impairment categorized in community-dwelling older adults with and without dementia using in-home sensors that recognise activities of daily living. Sci Rep. 2017 Feb 8;7:42084. doi: 10.1038/srep42084. PMID 28176828
- [Background] Wimo A, Jonsson L, Bond J, Prince M, Winblad B; Alzheimer Disease International. The worldwide economic impact of dementia 2010. Alzheimers Dement. 2013 Jan;9(1):1-11.e3. doi: 10.1016/j.jalz.2012.11.006. PMID 23305821